CLINICAL TRIAL: NCT04122040
Title: Effects of Roxithromycin on Quality of Life and Physiologic Outcomes in Bronchiectasis Patients During Treatment and Posttreatment Period
Brief Title: Effects of Roxithromycin on Quality of Life and Physiological Outcomes in Bronchiectasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Siwasak Juthong, Faculty of Medicine, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 54-282-14-3-2
Record Dates: First submitted 2019-10-08; First posted 2019-10-10 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Quality of Life; Respiratory Function Tests
Keywords: Bronchiectasis; quality of life; pulmonary function tests
MeSH Terms: conditions — Bronchiectasis | interventions — Roxithromycin

STUDY DESIGN:
Intervention Model Description: randomised control study
Who Masked: Investigator
Masking Description: block of 4
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- roxithromycin (Active Comparator): roxithromycin 300 mg oral per day
  Interventions: Drug: Roxithromycin 300 MG
- placebo (Placebo Comparator): placebo one tablet per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Roxithromycin 300 MG — Roxithromycin 300 mg oral per day
  Other Names: Roxithromycin
  Arms: roxithromycin
Drug: Placebo — Placebo one table oral once dialy
  Arms: placebo

SUMMARY:
roxithormycin 300 mg per day for 12 weeks could improve quality of life and physiological outcomes in bronchiectasis

DETAILED DESCRIPTION:
A randomized, double blinded, placebo controlled study was conducted to evaluate the effects of a 12-week administration of roxithromycin 300 mg once daily and a 12-week follow-up period in symptomatic stable bronchiectasis

ELIGIBILITY:
minimum 15 year maximum 75 years

Criteria inclusion Criteria:

Symptomatic bronchiectasis Stable clinical bronchiectasis

Exclusion Criteria:

Adverse drug reaction to macrolide Recent exacerbation within 2 weeks History of macrolide therapy within 2 weeks active malignancy and end stage diseases 5. not perform lung function tests Females who were lactating

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-03-01 (Actual); Primary Completion 2011-09-30 (Actual); Study Completion 2011-09-30 (Actual)

PRIMARY OUTCOMES:
SGRQ scores | for 12 weeks
  SGRQ scores

SECONDARY OUTCOMES:
pulmonary function tests | 24 weeks
  FEV1
sputum volumes | 24 wekse
  sputum volume per day

CONTACTS AND LOCATIONS:
Overall Officials: Kanung Saejiam, MS, Study Director — Prince of Songkla University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nakamura H, Fujishima S, Inoue T, Ohkubo Y, Soejima K, Waki Y, Mori M, Urano T, Sakamaki F, Tasaka S, Ishizaka A, Kanazawa M, Yamaguchi K. Clinical and immunoregulatory effects of roxithromycin therapy for chronic respiratory tract infection. Eur Respir J. 1999 Jun;13(6):1371-9. doi: 10.1183/09031936.99.13613809. PMID 10445614